CLINICAL TRIAL: NCT02519842
Title: A Phase III, Randomized, Placebo-Controlled Clinical Trial to Study the Efficacy and Safety of MK-0517/Fosaprepitant and Ondansetron Versus Ondansetron for the Prevention of Chemotherapy-Induced Nausea and Vomiting (CINV) in Pediatric Subjects Receiving Emetogenic Chemotherapy
Brief Title: Efficacy and Safety Study of Fosaprepitant (MK-0517) Plus Ondansetron Versus Ondansetron Alone for the Prevention of Chemotherapy-Induced Nausea and Vomiting in Pediatric Participants (MK-0517-044)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Further data are no longer required to support an application for use in pediatric patients. The decision to terminate was not based on any new safety findings
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0517-044; 2014-001783-34 (EudraCT Number); MK-0517-044 (Other: Merck Protocol Number)
Record Dates: First submitted 2015-08-07; First posted 2015-08-11 (Estimated); Results first posted 2018-03-08 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — fosaprepitant; Ondansetron; Dexamethasone; Serotonin 5-HT3 Receptor Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Fosaprepitant Regimen Cycle 1 (Experimental): Participants received a single dose of fosaprepitant 150 mg (or age-based adjustment) administered intravenously (IV) on Day 1 prior to chemotherapy plus ondansetron IV on Day 1 prior to chemotherapy and at investigator's discretion on day(s) of chemotherapy and up to 24 hours after chemotherapy. Participants may have also received dexamethasone IV at investigator's discretion on day(s) of chemotherapy and up to 24 hours after chemotherapy.
  Interventions: Drug: Fosaprepitant; Drug: Ondansetron; Drug: Dexamethasone
- Control Regimen Cycle 1 (Placebo Comparator): Participants received a single dose of matched placebo for fosaprepitant IV on Day 1 prior to chemotherapy plus ondansetron IV on Day 1 prior to chemotherapy and at investigator's discretion on day(s) of chemotherapy and up to 24 hours after chemotherapy. Participants may have also received dexamethasone IV at investigator's discretion on day(s) of chemotherapy and up to 24 hours after chemotherapy.
  Interventions: Drug: Placebo for fosaprepitant; Drug: Ondansetron; Drug: Dexamethasone
- Fosaprepitant Regimen Cycles 2-6 (Experimental): Participants received a single dose of fosaprepitant 150 mg (or age-based adjustment) IV on Day 1 prior to chemotherapy plus a 5-hydroxytryptamine 3 (5-HT3) antagonist on Day 1 prior to chemotherapy and per product label or standard of care. Participants may also have received dexamethasone IV at investigator's discretion on day(s) of chemotherapy and up to 24 hours after chemotherapy.
  Interventions: Drug: Fosaprepitant; Drug: Dexamethasone; Drug: 5-HT3 antagonist

INTERVENTIONS:
Drug: Fosaprepitant
  Other Names: EMEND for injection®
  Arms: Fosaprepitant Regimen Cycle 1; Fosaprepitant Regimen Cycles 2-6
Drug: Placebo for fosaprepitant
  Arms: Control Regimen Cycle 1
Drug: Ondansetron
  Other Names: Zofran®
  Arms: Control Regimen Cycle 1; Fosaprepitant Regimen Cycle 1
Drug: Dexamethasone
Drug: 5-HT3 antagonist
  Arms: Fosaprepitant Regimen Cycles 2-6

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of fosaprepitant (MK-0517) plus ondansetron versus ondansetron alone for the prevention of chemotherapy-induced nausea and vomiting (CINV) in pediatric participants scheduled to receive chemotherapeutic agent(s) associated with moderate or high risk of causing emesis (vomiting), or chemotherapy agent(s) not previously tolerated due to vomiting. The primary hypothesis is that a single dose of fosaprepitant in combination with ondansetron provides superior control of CINV compared to ondansetron alone as measured by the percentage of participants with a Complete Response (no vomiting, no retching, and no use of rescue medications) in the delayed phase (>24 to 120 hours) following initiation of emetogneic chemotherapy in Cycle 1.

DETAILED DESCRIPTION:
In Cycle 1, participants will receive double-blind study drug (fosaprepitant plus ondansetron with or without dexamethasone OR placebo to fosaprepitant plus ondansetron with or without dexamethasone). Upon completion of Cycle 1, participants may have the option to continue for up to 5 additional open-label cycles, receiving fosaprepitant plus ondansetron with or without dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* Is 0 (at least 37 weeks gestation) to 17 years of age at time of randomization
* Has a Lansky Play Performance score ≥60 (participants ≤16 years of age) or a Karnofsky score ≥60 (participants >16 years of age)
* Has a predicted life expectancy ≥3 months
* Is receiving chemotherapeutic agent(s) associated with moderate or high risk of emetogenicity, or a chemotherapy regimen not previously tolerated due to vomiting
* Has a preexisting functional central venous catheter available for study drug administration
* Is male OR is female who is not of reproductive potential OR is female who is of reproductive potential and agrees to avoid becoming pregnant in the 28 days prior to receiving study drug, while receiving study drug and for at least 30 days after last dose of study drug

Exclusion Criteria:

* Has vomited in the 24 hours prior to chemotherapy initiation on Treatment Day 1
* Has a symptomatic primary or metastatic central nervous system (CNS) malignancy with nausea and/or vomiting (asymptomatic participants may participate in study)
* Will be receiving stem cell rescue therapy in conjunction with study-related course of emetogenic chemotherapy or during the 14 days following administration of fosaprepitant/placebo for fosaprepitant
* Has received or will receive total body irradiation of radiation therapy to the abdomen or pelvis in the week prior to Treatment Day 1 and/or during the diary reporting period (120 hours following initiation of chemotherapy)
* Has had benzodiazepine, opioid or opioid like therapy initiated within 48 hours prior to study drug administration, or is expected to receive within 120 hours following initiation of chemotherapy except for single doses of midazolam, temazepam or triazolam
* Has started on systemic corticosteroid therapy within 72 hours prior to study drug administration or is expected to receive a corticosteroid as part of the chemotherapy regimen
* Is currently taking, or has taken within 48 hours of Treatment Day 1 the following drugs with antiemetic properties: 5-hydroxytryptamine 3 (5-HT3) antagonists (e.g., ondansetron), benzamides (e.g., haloperidol), cyclizine, domperidone, herbal therapies with potential antiemetic properties, olanzapine, phenothiazines (e.g., prochlorpenzine), scopolamine (this is not an exhaustive list)
* Is or has an immediate family member who is investigational site or sponsor staff directly involved with this study
* Is currently a user of any recreational or illicit drugs (including marijuana) or has current evidence of drug or alcohol abuse or dependence
* Is mentally incapacitated or has a significant emotional or psychiatric disorder
* Is pregnant or breast feeding
* Is allergic to fosaprepitant, aprepitant (MK-0869), ondansetron, or any other 5-HT3 antagonist
* Has a known history of QT prolongation or is taking any medication that is known to lead to QT prolongation
* Has an active infection (e.g., pneumonia), congestive heart failure, bradyarrhythmia, any uncontrolled disease (e.g., diabetic ketoacidosis, gastrointestinal obstruction) except for malignancy
* Has ever participated in a previous study of aprepitant or fosaprepitant or has taken an investigational drug with the last 4 weeks.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2017-02-24 (Actual); Study Completion 2017-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants for chemotherapy Cycles 1-6 were 0-17 years old and had documented malignancies and were scheduled to receive chemotherapeutic agent(s) associated with moderate or high risk of emetogenicity. Participants entering Cycles 2-6 must have completed Cycle 1 and had no unresolved drug-related adverse events.
Pre-assignment Details: Participants received double-blinded fosaprepitant+ondansetron with/without dexamethasone OR placebo + ondansetron with/without dexamethasone in Cycle 1. Upon completion of Cycle 1, participants from both Cycle 1 arms had the option to continue for 5 cycles of open-label fosaprepitant + 5-hydroxytryptamine 3 antagonist with/without dexamethasone.
Period: Base Study: Cycle 1
Arm/Group | Fosaprepitant Regimen Cycle 1 | Control Regimen Cycle 1 | Fosaprepitant Regimen Cycles 2-6
Started | 38 (Participants who completed Cycle 1 were invited to participate in optional Cycles 2-6.) | 37 (Participants who completed Cycle 1 were invited to participate in optional Cycles 2-6.) | 0
Treated | 37 | 34 | 0
Completed | 36 | 34 | 0
Not Completed | 2 | 3 | 0
Not completed — Screening Failure | 1 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawn by Parent/Guardian | 0 | 1 | 0
Not completed — Non-compliance with Study Drug | 0 | 1 | 0
Period: Optional Extension: Cycles 2-6
Arm/Group | Fosaprepitant Regimen Cycle 1 | Control Regimen Cycle 1 | Fosaprepitant Regimen Cycles 2-6
Started | 0 (27 participants from this arm in Cycle 1 entered optional Cycles 2-6) | 0 (28 participants from this arm in Cycle 1 entered optional Cycles 2-6) | 55 (Enrollment in Cycles 2-6 was optional.)
Treated | 0 | 0 | 55
Completed | 0 | 0 | 26
Not Completed | 0 | 0 | 29
Not completed — Physician Decision | 0 | 0 | 5
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Withdrawal by Parent/Guardian | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1
Not completed — Did Not Respond to Chemotherapy | 0 | 0 | 2
Not completed — Completed Chemotherapy | 0 | 0 | 13
Not completed — Enrollment Terminated at Site | 0 | 0 | 1
Not completed — Cycle Eligibility Criteria Not Met | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Cycle 1 is the base study. The participants who completed Cycle 1 were invited to participate in optional Cycles 2-6; there were no new participants enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fosaprepitant Regimen Cycle 1 | Control Regimen Cycle 1 | Total
Number analyzed (Participants) | 38 | 37 | 75
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.8 (4.2) | 10.9 (4.4) | 10.9 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 24 | 21 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 8 | 6 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 28 | 28 | 56
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced a Complete Response During the Delayed Phase (>24 to 120 Hours Post Initiation of Chemotherapy) in Cycle 1
Description: Complete Response was defined as no vomiting, no retching, and no use of rescue medication following the initiation of emetogenic chemotherapy in Cycle 1. A vomiting episode was specified as one or more episodes of emesis (expulsion of stomach contents through the mouth) or retching/dry heaves (an attempt to vomit that is not productive of stomach contents). Distinct vomiting episodes were separated by the absence of emesis and retching for at least one minute. The date and time of each vomiting episode was recorded by participants in diaries at the time of occurrence. The percentage of participants with no vomiting and no retching episodes in the delayed phase, defined as the time period of >24 to120 hours post initiation of chemotherapy in Cycle 1, was calculated.
Time Frame: >24 to 120 hours post initiation of chemotherapy (1 to 15 days after the dose of study drug)
Population: All participants who received at least 1 dose of study drug during Cycle 1.
Measure: Number; unit: Percentage of Participants
Arm/Group | Fosaprepitant Regimen Cycle 1 | Control Regimen Cycle 1
Number analyzed (Participants) | 37 | 34
Percentage of Participants | 48.6 | 41.2

2. Primary Outcome: Percentage of Participants Who Experienced One or More Adverse Events
Description: An adverse event (AE) is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not it is considered related to the study drug. A statistical analysis was performed for Tier 2 AEs in Cycle 1 to compare the percentage of participants who received fosaprepitant regimen and experienced at least 1 Tier 2 AE compared with the percentage of participants in the control regimen. The Tier 2 endpoint included broad clinical and laboratory AE categories consisting of the percentage of participants with any AE, drug-related AE, serious AE, and AEs that are both drug-related and serious. Tier 2 AEs were not pre-specified as events of interest and inclusion in the Tier 2 analysis required that at least 4 participants in any treatment group exhibited the AE.
Time Frame: Up to 6.5 months (up to 2 weeks after last dose of study drug)
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Groups:
- Fosaprepitant Regimen Cycles 2-6: Participants received a single dose of fosaprepitant 150 mg (or age-based adjustment) IV on Day 1 prior to chemotherapy plus a 5-HT3 antagonist on Day 1 prior to chemotherapy and per product label or standard of care. Participants may also have received dexamethasone IV at investigator's discretion on day(s) of chemotherapy and up to 24 hours after chemotherapy.
Arm/Group | Fosaprepitant Regimen Cycle 1 | Control Regimen Cycle 1 | Fosaprepitant Regimen Cycles 2-6
Number analyzed (Participants) | 37 | 34 | 55
Percentage of Participants | 89.2 | 79.4 | 78.2
Statistical Analysis 1: Comparison: Fosaprepitant Regimen Cycle 1 vs Control Regimen Cycle 1; Test type: Other; Mean Difference (Final Values) = 9.8, 95% CI 2-sided [-7.6 to 27.9] — Mean difference in percentage of participants who experienced at least 1 tier 2 AE and received fosaprepitant regimen compared with participants who received control regimen

3. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not it is considered related to the study drug. A statistical analysis was performed to compare the percentage of participants who discontinued in Cycle 1 due to an AE and received fosaprepitant regimen compared with the percentage of participants who received control regimen.
Time Frame: Up to 6 months (up to last dose of study drug)
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Fosaprepitant Regimen Cycle 1 | Control Regimen Cycle 1 | Fosaprepitant Regimen Cycles 2-6
Number analyzed (Participants) | 37 | 34 | 55
Percentage of Participants | 5.4 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Fosaprepitant Regimen Cycle 1 vs Control Regimen Cycle 1; Test type: Other; Mean Difference (Final Values) = 5.4, 95% CI 2-sided [-5.1 to 17.8] — Mean difference in percentage of participants who discontinued due to an AE and received fosaprepitant regimen compared with participants who received control regimen

4. Secondary Outcome: Percentage of Participants Who Experienced a Complete Response During the Acute Phase (0 to 24 Hours Post Initiation of Chemotherapy) in Cycle 1
Description: Complete Response was defined as no vomiting, no retching, and no use of rescue medication following the initiation of emetogenic chemotherapy in Cycle 1. A vomiting episode was specified as one or more episodes of emesis (expulsion of stomach contents through the mouth) or retching/dry heaves (an attempt to vomit that is not productive of stomach contents). Distinct vomiting episodes were separated by the absence of emesis and retching for at least one minute. The date and time of each vomiting episode was recorded by participants in diaries at the time of occurrence. The percentage of participants with no vomiting and no retching episodes in the acute phase, defined as the time period of 0 to 24 hours post initiation of chemotherapy in Cycle 1, was calculated.
Time Frame: 0 to 24 hours post initiation of chemotherapy (up to 1 day after the dose of study drug)
Population: All participants who received at least 1 dose of study drug during Cycle 1.
Measure: Number; unit: Percentage of Participants
Arm/Group | Fosaprepitant Regimen Cycle 1 | Control Regimen Cycle 1
Number analyzed (Participants) | 37 | 34
Percentage of Participants | 70.3 | 58.8

5. Secondary Outcome: Percentage of Participants Who Experienced a Complete Response During the Overall Phase (0 to 120 Hours Post Initiation of Chemotherapy) in Cycle 1
Description: Complete Response was defined as no vomiting, no retching, and no use of rescue medication following the initiation of emetogenic chemotherapy in Cycle 1. A vomiting episode was specified as one or more episodes of emesis (expulsion of stomach contents through the mouth) or retching/dry heaves (an attempt to vomit that is not productive of stomach contents). Distinct vomiting episodes were separated by the absence of emesis and retching for at least one minute. The date and time of each vomiting episode was recorded by participants in diaries at the time of occurrence. The percentage of participants with no vomiting and no retching episodes in the overall phase, defined as the time period of 0 to 120 hours post initiation of chemotherapy in Cycle 1, was calculated.
Time Frame: 0 to 120 hours post initiation of chemotherapy (up to 15 days after the dose of study drug)
Population: All participants who received at least 1 dose of study drug during Cycle 1.
Measure: Number; unit: Percentage of Participants
Arm/Group | Fosaprepitant Regimen Cycle 1 | Control Regimen Cycle 1
Number analyzed (Participants) | 37 | 34
Percentage of Participants | 40.5 | 32.4

6. Secondary Outcome: Percentage of Participants Who Experienced No Vomiting, Regardless of Rescue Medication Use, During the Overall Phase (0 to 120 Hours Post Initiation of Chemotherapy) in Cycle 1
Description: Vomiting was assessed, regardless of rescue medicine use, following the initiation of emetogenic chemotherapy in Cycle 1. A vomiting episode was specified as one or more episodes of emesis (expulsion of stomach contents through the mouth) or retching/dry heaves (an attempt to vomit that is not productive of stomach contents). Distinct vomiting episodes were separated by the absence of emesis and retching for at least one minute. The date and time of each vomiting episode was recorded by participants in diaries at the time of occurrence. Rescue medication was permitted to alleviate symptoms of established nausea or vomiting; but not as preventive medication. The percentage of participants with no vomiting and no retching episodes in the overall phase, defined as the time period of 0 to 120 hours post initiation of chemotherapy in Cycle 1, was calculated.
Time Frame: 0 to 120 hours post initiation of chemotherapy (up to 15 days after the dose of study drug)
Population: All participants who received at least 1 dose of study drug during Cycle 1.
Measure: Number; unit: Percentage of Participants
Arm/Group | Fosaprepitant Regimen Cycle 1 | Control Regimen Cycle 1
Number analyzed (Participants) | 37 | 34
Percentage of Participants | 40.5 | 32.4

ADVERSE EVENTS:
Time Frame: Adverse events data were collected up to 6.5 months (from start of study drug and up to 14 days after the last dose for each cycle in Cycles 1-6).
Description: This safety analysis was based on all participants who received at least 1 dose of study drug during Cycles 1 through 6. Cycle 1 is the base study. The participants who completed Cycle 1 were invited to participate in optional Cycles 2-6; there were no new participants enrolled.
Arm/Group | Fosaprepitant Regimen Cycle 1 | Control Regimen Cycle 1 | Fosaprepitant Regimen Cycles 2-6
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/34 | 1/55
Serious Adverse Events (participants affected / at risk) | 11/37 | 8/34 | 28/55
Other Adverse Events (participants affected / at risk) | 28/37 | 18/34 | 30/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosaprepitant Regimen Cycle 1 (N=37) | Control Regimen Cycle 1 (N=34) | Fosaprepitant Regimen Cycles 2-6 (N=55)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (3)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 3 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 5 (5) | 19 (32)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Soft tissue inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media chronic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diet refusal (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Thrombosis in device (Product Issues) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosaprepitant Regimen Cycle 1 (N=37) | Control Regimen Cycle 1 (N=34) | Fosaprepitant Regimen Cycles 2-6 (N=55)
Anaemia (Blood and lymphatic system disorders) | 11 (11) | 3 (3) | 11 (20)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0) | 7 (15)
Neutropenia (Blood and lymphatic system disorders) | 5 (6) | 3 (3) | 4 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (8) | 2 (2) | 7 (14)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 1 (1) | 6 (9)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (3) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 9 (14)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1) | 11 (24)
Fatigue (General disorders) | 0 (0) | 2 (2) | 1 (2)
Mucosal inflammation (General disorders) | 3 (4) | 0 (0) | 4 (6)
Pyrexia (General disorders) | 4 (5) | 0 (0) | 7 (8)
Alanine aminotransferase increased (Investigations) | 2 (2) | 3 (3) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 2 (3)
Neutrophil count decreased (Investigations) | 6 (6) | 3 (3) | 2 (2)
Platelet count decreased (Investigations) | 4 (4) | 3 (5) | 5 (32)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrollment was terminated early because the data were not necessary to support a claim in pediatric participants and not due to safety concerns. The last participant enrolled on 2016-08-05 and enrolled participants were active until study completion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT02519842/Prot_SAP_000.pdf